CLINICAL TRIAL: NCT03601572
Title: Hypnoanalgesia in Surgical and Endovenous Treatment of Varicosis
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned research
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0453
Record Dates: First submitted 2018-01-11; First posted 2018-07-26 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2017-12

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Endoveinous treatment of saphenous varicoses and phlebectomia of tributary veins are commonly performed under local anesthesia. Hypnoanalgesia might reduce perinterventional pain.

This study has the aim to test the effectiveness of hypnoanalgesia, performed by a specialised nurse, for peri-and post-procedual pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* patients treated under local anesthesia by Laser or radiofrequency or phlebectomies for their varicose veins
* Age of 18 and over

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients treated under local anesthesia by Laser or radiofrequency or phlebectomies for their varicose veins
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of hypnosis | on intraoperative
  Assessment of the contribution of hypnosis in patients who will be treated under local anesthesia by Laser or radiofrequency or phlebectomies for their varicose veins
Evaluate the effects of hypnosis | 1 day
  Assessment of the contribution of hypnosis in patients who will be treated under local anesthesia by Laser or radiofrequency or phlebectomies for their varicose veins

CONTACTS AND LOCATIONS:
Overall Officials: GUDRUN BOGE, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC